CLINICAL TRIAL: NCT02190539
Title: The Banerji Protocol for Advanced Breast Cancer- Feasibility Study
Brief Title: Homeopathic Protocol for Advanced Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to recruit patients
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Moshe Frenkel, MD, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0050-14-MMC
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; complementary medicine; homeopathy; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Homeopathic treatment (Experimental): A feasibility study examining whether patients with advanced breast cancer would follow a homeopathic protocol for three to six months.
  Interventions: Other: Homeopathic treatment

INTERVENTIONS:
Other: Homeopathic treatment — Remedies are sold over the counter without a physician prescription (approved by the Israeli Ministry of Health). No toxicity or side effects are expected to be observed, potencies (dilutions) of substances beyond 7C (7 dilutions, each 1:100) do not contain a sufficient number of molecules of the original material to be pharmacologically active. Since the remedies being used in this trial are diluted at 30c and 200c, levels that are way beyond Avogrado's number, so no original material is expected to be found. This fact was verified utilizing high pressure liquid chromatography (HPLC) method. Due to those facts, most scientists do not accept that these remedies have any biological effects and consign any positive response to the placebo effect.
  Other Names: A combined treatment of three homeopathic remedies:; Phytolacca 200C; Thuja 30C; Carcinosin 30c

SUMMARY:
The objective of this study is to conduct a feasibility study at Meir Oncology Institute examining whether patients with advanced breast cancer would follow a homeopathic protocol for three to six months.

The primary aim of the study is to establish if patients with advanced breast cancer in Meir Oncology Institute would follow a regimen of treatment as used by Dr Banerji in India, for six months.

The secondary aim is to observe the quality of life and wellbeing of patients undergoing this protocol

DETAILED DESCRIPTION:
- Homeopathy is a controversial system of care and at the center of the controversy lays the question of whether high dilution remedies can be effective.

There have been only a handful of high quality studies of homeopathy on the treatment of cancer, despite its widespread use for this condition.

In a recent prospective observational study done in Germany with cancer patients in two differently treated cohorts it was observed that an improvement in quality of life was observed in patients taking the addition of homeopathic treatment. In the laboratory, research on homeopathy and cancer that does exist is limited but has some clues for effects that cannot be ignored. A study that was conducted at The University of Texas MD Anderson Cancer Center, revealed that four ultradilute remedies (Carcinosin, Phytolacca, Conium, and Thuja) exerted preferential cytotoxic effects against two breast cancer cell lines, causing cell cycle delay/arrest and apoptosis without affecting the normal mammary epithelial cells. Since patients with advanced breast cancer are the highest CAM users amongst patients affected by cancer, it was thought that a feasibility study with this group of patients, would be a rational first step in proceeding to evaluate this controversial method of care, if it has merit or not.

* The objective of this study is to conduct a feasibility study at Meir Oncology Institute examining whether patients with advanced breast cancer would follow a homeopathic protocol for three to six months. The primary aim of the study is to establish if patients with advanced breast cancer in Meir Oncology Institute would follow homeopathic protocol as used by Dr Banerji in India, for six months. The secondary aim is to observe the quality of life and wellbeing of patients undergoing this protocol.
* Patients with the diagnosis of advanced breast cancer who attend the Meir Oncology Institute clinic will be offered by their treating physician or nurse a fact sheet about this study and will be asked to participate in this protocol. The protocol will be explained to the patient by the research team. If they agree to participate they will be given a consent form to sign, and basic information will be obtained from each patient. This information will include basic demographics (age, marital status, employment , education level) and basic medical information ( Disease status and progress, current symptoms, medications and treatments being used, complementary medicine being used) as well as evaluation of quality of life using the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ).
* Patients will receive the selected homeopathic remedies (Carcinosin 30C, Phytolacca 200C, and Thuja 30C) with written instructions about the proper use of the remedies. The remedies will be offered to patients in addition to their regular conventional care. Patients that cannot participate in conventional cancer care due to side effects, expected adverse reactions or other reasons that prevent them from utilizing conventional care will be offered to participate in the study, as well. In addition, patients who for their own reasons elect to refuse conventional treatment can be offered to participate in the study in order to keep them in the system and not lose them to alternative untested treatments. Every 4 weeks for the period of 3 months and once at 6 months, a research assistant/ research nurse will contact each participant to review EORTC QLQ- C-30 questionnaire to evaluate quality of life as well as a follow up questionnaire which will verify the actual use of these remedies, perceived problems in taking these remedies, utilization of other therapies, address patients concerns, and document disease progression. A total of 30 patients will be enrolled in this study and their data will be reviewed and analyzed six months after recruitment to the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to speak and read Hebrew/English with patients residing in Israel.
* Diagnosis of advanced breast cancer treated and followed in Meir Oncology Institute
* Patients that cannot participate in conventional cancer care due to side effects, expected adverse reactions or other reasons that prevent them from utilizing conventional care.
* Patients, who for their own reasons elect to refuse conventional treatment, can be offered to participate in the study in order to keep them in the system and not lose them to alternative untested treatments.
* Consent to participate in this study

Exclusion Criteria:

* Inability to understand the intent of the study and follow the instructions
* Medical condition that would preclude participation in an interview session lasting 15-30 minutes
* Diagnosis of active psychosis or severe cognitive impairment confirmed by the patient's attending physician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
To establish if patients with advanced breast cancer in Meir Oncology Institute would follow a homeopathic treatment protocol as used by Dr Banerji in India, for six months. | Six months
  Investigators will follow patients with advanced breast cancer in Meir Oncology Institute and see if patients would follow a homeopathic treatment protocol as used by Dr Banerji in India, for six months.

SECONDARY OUTCOMES:
Observe and verify the quality of life and wellbeing of patients undergoing this protocol | Six months
  Investigators will document the quality of life and wellbeing of patients undergoing this protocol utilizing the EORTC QLQ-C30 (a questionnaire developed to assess the quality of life of cancer patients).

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Frenkel, MD, Principal Investigator — Institute of Oncology Meir Medical Center
Locations (1):
- Institute of Oncology Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Yes
Publications, Presentations in international meetings

REFERENCES:
- [Result] Frenkel M, Mishra BM, Sen S, Yang P, Pawlus A, Vence L, Leblanc A, Cohen L, Banerji P, Banerji P. Cytotoxic effects of ultra-diluted remedies on breast cancer cells. Int J Oncol. 2010 Feb;36(2):395-403. PMID 20043074
- See also: Integrative Oncology - Homeopathy — http://www.moshefrenkelmd.com/index.asp?page=2171&lang=eng